CLINICAL TRIAL: NCT06727552
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Barzolvolimab in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Barzolvolimab in Patients With Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-15
Record Dates: First submitted 2024-12-09; First posted 2024-12-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: AD; Atopic Dermatitis; eczema; barzolvolimab; CDX-0159; CDX0159-15
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Barzolvolimab 150 mg (Experimental): Barzolvolimab loading dose of 450 mg subcutaneous injection followed by 150 mg administered every 4 weeks for 32 weeks
  Interventions: Biological: Barzolvolimab
- Barzolvolimab 300 mg (Experimental): Barzolvolimab loading dose of 450 mg subcutaneous injection followed by 300 mg administered every 4 weeks for 32 weeks
  Interventions: Biological: Barzolvolimab
- Placebo then barzolvolimab 150 mg (Experimental): Placebo subcutaneous injection every 4 weeks for 16 weeks and then barzolvolimab loading dose of 450 mg followed by 150 mg administered every 4 weeks for 16 weeks.
  Interventions: Biological: Barzolvolimab; Drug: Matching placebo
- Placebo then barzolvolimab 300 mg (Experimental): Placebo subcutaneous injection every 4 weeks for 16 weeks and then barzolvolimab loading dose of 450 mg followed by 300 mg administered every 4 weeks for 16 weeks.
  Interventions: Biological: Barzolvolimab; Drug: Matching placebo

INTERVENTIONS:
Biological: Barzolvolimab — Subcutaneous Administration
Drug: Matching placebo — Subcutaneous Administration
  Arms: Placebo then barzolvolimab 150 mg; Placebo then barzolvolimab 300 mg

SUMMARY:
The purpose of this study is to assess the efficacy and safety of barzolvolimab in adults with Atopic Dermatitis

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel group, placebo controlled phase 2 study to assess the efficacy and safety of barzolvolimab (CDX-0159) in adult participants with Atopic Dermatitis.

There is a screening period of up to 28 days, a 16-week double-blind, placebo-controlled treatment period, a 16-week double-blind, active treatment period, and a 16-week follow-up period. On Day 1, participants will be randomly assigned on a 1:1:1 ratio to receive barzolvolimab (CDX-0159) by subcutaneous injections of 150 mg every 4 weeks (Q4W) after an initial loading dose of 450 mg [Arm 1], 300 mg Q4W after an initial loading dose of 450 mg [Arm 2], or placebo Q4W [Arm 3]. At Week 16, participants on placebo will be re-randomized on a 1:1 ratio to receive barzolvolimab by subcutaneous injections of 150 mg every 4 weeks (Q4W) after an initial loading dose of 450 mg, 300 mg Q4W after an initial loading dose of 450 mg. Participants on Arms 1 and 2 will undergo a mock re-randomization at Week 16 to maintain the blind.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Diagnosis of chronic atopic dermatitis (AD) for at least 1 year
3. Onset of symptoms at least 1 year prior and current symptoms consistent with moderate to severe AD as defined by:

   1. EASI ≥ 12 at Visit 1 and EASI ≥ 16 at Visit 2
   2. Body Surface Area of Involvement (BSA) ≥ 10% at Visit 1 and Visit 2
   3. IGA score ≥ 3 at Visit 1 and Visit 2
   4. Severe itch, defined by weekly average of daily PP-NRS score of ≥ 5, during the 7 days prior to treatment
4. Documented history of inadequate response to treatment with topical medications or for whom topical medications are otherwise medically inadvisable.
5. Willing and able to complete a daily symptom electronic diary for the duration of the study and adhere to the study visit schedule.

Exclusion Criteria:

1. Any other active pruritic skin diseases that would confound AD assessments based on the Investigator's clinical judgment.
2. Phototherapy with ultraviolet (UV) A or UVB within 4 weeks of Visit 1.
3. Planned or anticipated use of any prohibited medications at any time during the study.
4. Prior receipt of barzolvolimab or other anti-KIT therapy. There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline in the weekly average of the daily Peak Pruritus Numerical Rating Scale (PP-NRS) score at Week 16 | From Day 1 (first dose) to Day 113 (week 16)
  Evaluate the clinical efficacy of 2 dose levels (150 mg and 300 mg) of barzolvolimab, compared to placebo, in adult participants with moderate to severe atopic dermatitis (AD) using the PP-NRS. The PP-NRS ranges from 0 = "no itch" to 10 ="worst imaginable itch" for the worst intensity itch in the preceding 24-hr period.

SECONDARY OUTCOMES:
Percent change from Baseline in Eczema Area Severity Index (EASI) score at Week 16. | From Day 1 (first dose) to Day 113 (week 16)
  A total EASI score range from 0 to 72 points will be recorded for each assessment, with higher scores reflecting worse severity of AD.
  * 0 = clear
  * 0.1-1.0 = almost clear
  * 1.1-7.0 = mild
  * 7.1-21.0 = moderate
  * 21.1-50.0 = severe
  * 50.1-72.0 = very severe
Proportion of participants achieving an Investigator Global Assessment (IGA) score of "0" or "1" at Week 16. | From Day 1 (first dose) to Day 113 (week 16)
  The IGA determines severity of AD and clinical response to treatment on a static 5-point scale based on erythema and papulation/infiltration
  * 0 = Clear
  * 1 = Almost clear
  * 2 = Mild
  * 3 = Moderate
  * 4 = Severe

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Cahaba Dermatology & Skin Health Center, LLC, Birmingham, Alabama
  - Ohara Aivaz MD Dermatology, Beverly Hills, California
  - Advanced Dermatology Center - Burbank, Burbank, California
  - 310 Clinical Research, Inglewood, California
  - Avance Trials, Laguna Niguel, California
  - LA Universal Research Center, Inc., Los Angeles, California
  - UCLA Division of Dermatology, Los Angeles, California
  - Dynasty Dermatology, Pasadena, California
  - Acclaim Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - FOMAT Medical Research - Allergy, Asthma, & Immunology Medical Group, Ventura, California
  - Pacific Clinical Innovations Inc., Vista, California
  - Focus Clinical Research, West Hills, California
  - Direct Helpers Research Center, Hialeah, Florida
  - University of Miami, Miami, Florida
  - International Dermatology Research Inc - Miami, Miami Lakes, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Well Pharma Medical Research Corporation, South Miami, Florida
  - Centricity Research Columbus Dermatology, Columbus, Georgia
  - Georgia Skin and Cancer Clinic, Savannah, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Center for Medical Dermatology + Immunology Research, Chicago, Illinois
  - Sneeze Wheeze and Itch Associates LLC, Normal, Illinois
  - Equity Medical LLC, Bowling Green, Kentucky
  - Allergy and Asthma Specialists PSC, Owensboro, Kentucky
  - Onyx Clinical Research - Michigan, Flint, Michigan
  - Derm Center, Troy, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Excel Clinical Research, Las Vegas, Nevada
  - Equity Medical, LLC, New York, New York
  - OptiSkin Medical, New York, New York
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Palmetto Clinical Trial Services LLC, Simpsonville, South Carolina
  - Zenos Clinical Research, Dallas, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Sienna Dermatology, Sugar Land, Texas
  - Center for Clinical Studies LTD.LLP, Webster, Texas
  - Jordan Valley Dermatology Center - South Jordan, South Jordan, Utah